CLINICAL TRIAL: NCT06991179
Title: A Phase 1, Open-Label Study to Evaluate the Effects of Food and Multiple-Doses of Esomeprazole on the Pharmacokinetics of a Single Oral Dose of LY4064809 in Healthy Adult Participants
Brief Title: A Study of Food Effect and Esomeprazole on LY4064809 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scorpion Therapeutics, a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27693; J6M-MC-JSGC (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-19; First posted 2025-05-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 Treatment A Fasted (Experimental): LY4064809 administered orally
  Interventions: Drug: LY4064809
- Group 1 Treatment B High-Fat Meal (Experimental): LY4064809 administered orally
  Interventions: Drug: LY4064809
- Group 2 Treatment A Fasted (Experimental): LY4064809 administered orally
  Interventions: Drug: LY4064809
- Group 2 Treatment C Proton Pump Inhibitor (PPI) Effect (Experimental): LY4064809 administered orally with esomeprazole
  Interventions: Drug: LY4064809

INTERVENTIONS:
Drug: LY4064809 — Administered orally

SUMMARY:
The purpose of this study is to evaluate the safety and effect of food on LY4064809 and the safety and effect of stomach changes by a proton pump inhibitor (PPI) esomeprazole, under fasted conditions in healthy adult participants. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy as determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations at screening and/or admission as assessed by the investigator (or designee)
* Participants have normal blood pressure and pulse rate, as determined by the investigator
* Have venous access sufficient to allow for blood sampling
* Have a body mass index (BMI) within the range 18-32 kilogram/square meter (kg/m²) (inclusive)
* Individuals not of childbearing potential and individuals assigned male at birth may participate in this trial

Exclusion Criteria:

* History or presence of any of the following conditions, deemed clinically significant by the investigator (or designee), which may significantly alter the absorption, metabolism, or elimination of drugs, constitute a risk when taking the study intervention or interfere with the data interpretation:

  * Metabolic disease, including congenital non-hemolytic hyperbilirubinemia (for example, Gilbert syndrome),
  * Biliary disease, including cholecystectomy,
  * Gastrointestinal (GI) disease,
  * Hematological disease,
  * Neurological disease,
  * Significant history of, or presence of hepatic disease, including any abnormal liver function tests and serum total bilirubin above the 1.5

    × upper limits of normal (ULN) range per the laboratory's reference ranges at screening or admission, or
  * Clinically significant, active cardiovascular disease or history of myocardial infarction within 6 months prior to the planned start of LY4064809
* History of a major surgical procedure within 30 days prior to screening
* Diagnosed and/or treated malignancy within 5 years prior to screening with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and curatively resected in situ carcinoma of the cervix.
* Have known allergies to LY4064809 or related compounds or esomeprazole or related compounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4064809 | Day 1 to Approximately Day 47
  PK: Cmax of LY4064809
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve from Time Zero to Time T (AUC 0-tlast) | Day 1 to Approximately Day 47
  PK: AUC 0-tlast, where t is the last time point with a measurable concentration
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve from Zero to Infinity (AUCinf) | Day 1 to Approximately Day 47
  PK: AUCinf

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLilly (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Pharmaron Clinical Pharmacology Center Inc, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No